CLINICAL TRIAL: NCT04634708
Title: The Use of the EXCOR Active Driving Unit for Mobilization of Pediatric Patients With Ventricular Assist Device Support
Acronym: E-Motion
Status: Completed | Type: Observational
Sponsor: Berlin Heart GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: E-20-330
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Heart Failure; Cardiomyopathies; Ventricular Dysfunction; Heart Diseases; Cardiovascular Diseases
Keywords: EXCOR Ventricular Assist Device; EXCOR Active; Mobilization; Pediatric
MeSH Terms: conditions — Heart Failure; Cardiomyopathies; Ventricular Dysfunction; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric patients on EXCOR VAD support
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention due to observational design

SUMMARY:
The purpose of this observational study is to evaluate the performance of the Berlin Heart EXCOR Active driving unit while being used with the approved EXCOR ventricular assist device system.

DETAILED DESCRIPTION:
The study has a prospective, multicenter, international, single arm, observational design.

Study enrollment is expected to take 18 months and subjects will be followed until they reach an outcome or for 45 days on the EXCOR Active driving unit. The overall study duration is expected to be approximately 20 months.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients meeting all indications as specified in the current version of the instructions for use (IFU) of the EXCOR® Active system,
* Age < 18 years,
* Patient and legal guardian has consented via signature on the study informed consent form,
* Patient is able to get mobilized according to hospital standard and is currently supported with the Ikus driving unit. The decision if a patient is able to get mobilized is at the discretion of the investigator.

Exclusion Criteria:

* Patient has any contraindication as specified in the current version of the IFU of the EXCOR® Active system,
* Patient and/or legal representative has not given written consent to participate in the study (non-consent),
* Females of childbearing age who are not on contraceptives or surgically sterile or who are pregnant.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Twenty patients supported with the EXCOR® VAD. Patients must meet the eligibility criteria as specified and must not meet the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
EXCOR Active device performance | 52 days

SECONDARY OUTCOMES:
Successful patient outcome rates | Whenever it happens or 52 days
  Successful outcome is defined as:
  * survival to transplant, or
  * survival to recovery/successful weaning, or
  * survival on EXCOR Pediatric at 45 days post-switch to EXCOR Active.

OTHER OUTCOMES:
Safety of the device | 52 days
  * Adverse Events and Adverse Device Effects
  * Serious Adverse Events and Serious Adverse Device Effects
Mobility | 52 days
  The mobility will be assessed with a patient diary.
Quality of Life of the Patient and Family | 52 days
  The QoL will be assessed with questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Deutsches Herzzentrum Berlin, Berlin, Germany